CLINICAL TRIAL: NCT06009328
Title: Correlation Between Fundamental Movement Skills, Body Mass Index, and Quality of Life in School Aged Children
Brief Title: Fundamental Movement Skills, Body Mass Index and Quality of Life in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Fahmy Hassan Al Nemr, lecturer in pediatric department, faculty of physical therapy, Cairo University
Other Study IDs: P.T.REC/012/003398
Record Dates: First submitted 2023-08-19; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Overweight Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: fundamental movement skills — measured by test of gross motor development

SUMMARY:
Early childhood obesity is a serious worldwide problem, and fundamental movement skills (FMS) are very important factors in human movement. Thus, several advanced studies have examined the associations between FMS, body mass index (BMI) and quality of life.

The purpose of this study was to investigate the relation between FMS, BMI and quality of life in Egyptian school aged children.

DETAILED DESCRIPTION:
A total of 216 primary school aged children, aged 5-7 y from both sex participated in this study. FMS were measured using the Test of Gross Motor Development-II (TGMD-II), and BMI was calculated as the weight (kg) divided by the square of the height (m) [weight/ height2] ,and quality of life was measured by PedsQol scale

ELIGIBILITY:
Inclusion Criteria:

- normal school aged children , aged 5-7 years with different weight categories

Exclusion Criteria:

* children with visual or auditory problems or those who experienced surgery in their lower limbs 1 year before study

Ages: 5 Years to 7 Years | Sex: All
Age Groups: Child
Study Population: normal school aged children from 5-8 years
Sampling Method: Non-Probability Sample
Enrollment: 216 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-11 (Estimated)

PRIMARY OUTCOMES:
test of gross motor development | 3 months
  a valid and reliable test for assessing fundamental movement skills in children aged 3-10 years
body mass index | 3 months
  used to assess anthropometric measurements
PedsQol scale | 3 months
  used to assess quality of life in children. generic core scale will be used and total score will be used in analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty Of Physical Therapy, Cairo, Egypt